CLINICAL TRIAL: NCT04866420
Title: The MenFAS Study: Understanding Mental Fatigue After Stroke
Brief Title: Understanding Mental Fatigue After Stroke
Acronym: MenFAS
Status: Completed | Type: Observational
Sponsor: Oxford Brookes University (Other)
Responsible Party: Principal Investigator, Avril Dillon, Elizabeth Casson Trust PhD Scholar, Oxford Brookes University
Other Study IDs: 201376
Record Dates: First submitted 2021-04-22; First posted 2021-04-29 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Post-Stroke Fatigue; Fatigue
Keywords: Cognitive impairment; Attention
MeSH Terms: conditions — Stroke; Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Poststroke fatigue: Participants who are experiencing fatigue post stroke.
  Interventions: Behavioral: The MenFAS Study

INTERVENTIONS:
Behavioral: The MenFAS Study — A cross over repeated exposure randomized design observational study

SUMMARY:
Mental fatigue is a major problem for stroke survivors and sometimes remains present years after the event. It is often rated as the most persisting and frustrating symptom. For many, mental fatigue has a significant negative effect on rehabilitation, and patients report difficulties with returning to previous levels of participation in their meaningful everyday activities whether at home, work or in the community.

The development of effective evidence based interventions have been limited by our understanding of post stroke fatigue. This may be attributed to the fact that the underlying mechanisms for post stroke mental fatigue are unknown. Evolving theories suggest that mental fatigue may be associated with a dysfunction in the cognitive domain of attention.

An impairment in the domain of attention may result in previously effortless activities of daily living that require sustained attention to become exhausting. Specific knowledge on the influence of background noise and other distractions on a person's ability to sustain attention after stroke is lacking. This research project will contribute to new and important knowledge in this area.

A total of 30 adults will be reviewed at least 2 months after stroke on tasks that require sustained attention. The investigators plan to observe the influence background distraction has on the ability to do these tasks and whether wearing earphones will assist with concentration levels, and reduce fatiguing situations.

This project provides a unique opportunity to investigate how a dysfunction in the cognitive domain of attention may be related to the experience of mental fatigue after stroke. The investigators will use a reaction time based test, fatigue questionnaires, alongside the wearing of earphones when examining associations. This knowledge may help to determine who is at risk of developing symptoms of mental fatigue. Furthermore, it may shed a light on possible prevention strategies, and provide more suitable guidance to those affected by mental fatigue.

DETAILED DESCRIPTION:
Fatigue is reported by stroke survivors as a highly problematic and persisting experience with many rating it as their most severe amongst all post - stroke sequelae. Given the negative impact of fatigue on participation, an investigation into the possible underlying mechanisms mediating fatigue after stroke has clinical implications.

Recent studies indicate that an impairment in the domain of attention is related to the experience of higher fatigue levels. However, the complexity of this mechanism, presentation and measurement have made the findings unclear. In studies, testing methods to identify a dysfunction in the domain of attention can be mentally fatiguing. Moreover, it is not clear whether the impact of contextual factors on concentration levels, such as background noise and distraction, has been considered.

Primary Objective:

Among people with stroke engaging in a task requiring sustained attention, to what extent does the use of noise-cancelling earphones impact on mental fatigue? Fatigue will be assessed using two measures: 1) The Continuous Performance Test, a reaction time based assessment completed on a computer tablet and 2) A Visual Analog Scale for Fatigue, which is paper based.

Design: A cross - over repeated exposure randomised design will be used. Study participants will be randomised to do tasks of sustained attention, followed by a reaction time based assessment on a tablet, first with and then without earphones or first without and then with earphones. The two assessment sessions will be done one week apart to allow for a washout period. Participants will be invited to rank their fatigue levels on a visual analog scale, pre - post these assessments.

Secondary Objectives:

* Is baseline cognitive fatigue a predictor for performance decrement on tasks of sustained attention? This will be assessed using the Fatigue Scale for Motor and Cognitive Functions (FSMC). This scale includes both physical and cognitive aspects of fatigue.
* What are the contextual factors mediating fatigue symptoms? This will be assessed using a momentary ecological assessment application on a mobile phone or a diary paper based assessment.
* What is the influence of fatigue symptoms on participatory patterns as seen on the ecological momentary app or diary? This will be assessed with a wrist worn Accelerometer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke
* Are over the age of 18 (no upper limit)
* Ability to understand spoken and / or written English

Exclusion Criteria:

* Not functionally able to undergo neuropsychological assessment or reply to questionnaires. This will be assessed on the cognitive screen, the Oxford Cognitive Screen (OCS).
* Medically unstable or have another condition that could impact results (e.g. substance abuse).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will be > 2 months post stroke and will be in this study for a maximum 4 week period, consisting of two sessions at home.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-12-05 (Actual); Study Completion 2021-12-05 (Actual)

PRIMARY OUTCOMES:
The Continuous Performance Task | 12 minutes
  The Continuous Performance Task (CPT) is a computerised reaction time test and is one of the most frequently used, objective tools to measure sustained attention over time. This assessment takes 12 minutes. Sustained attention will be assessed based on changes on performance over time. The task will be completed twice (once with, once without earphones) over the two assessment days.
Change in baseline fatigue at 2 hours - Visual Analog Scale for fatigue | 4 x across 2 testing days (1 week apart). Day 1: Before (baseline) and after reaction time assessment (2hours). Day 2: Before (baseline) and after reaction time assessment (2hours)
  A VAS consisting of a 10cm vertical line from 1 (no fatigue) to 10 (worst possible fatigue) will be used to obtain the momentary fatigue associated with completing the task of sustained attention. Participants will rank their mental fatigue at the beginning and the end of each reaction time task (on the CPT) performed.

SECONDARY OUTCOMES:
Fatigue Scale for Motor and Cognitive functions. | Baseline fatigue.
  Baseline fatigue will be measured using the self-reported Fatigue Scale for Motor and Cognitive Functions (FSMC) which has been validated for use in neurological conditions, including stroke (Ref -Hubs). This scale includes both physical and cognitive fatigue. Cut-off values for the FSMC total scale and both subscales were determined by standard deviations from the mean values of healthy control population in two other studies (Hubacher et al 2012; Penner et al 2009). Subdivision from mild, moderate to severe fatigue for both domains as well as for the composite fatigue score are provided:
  FSMC Sum Score ≥43 Mild fatigue, ≥53 Moderate fatigue, ≥63 Severe fatigue. FSMC Cognitive Score ≥22 Mild cognitive fatigue ≥ 28 Moderate cognitive fatigue ≥ 34 Severe cognitive fatigue FSMC Physical Score ≥ 22 Mild motor fatigue, ≥27 Moderate motor fatigue, ≥32 Severe motor fatigue.
Oxford Cognitive Screen | Baseline cognitive abilities
  Baseline cognitive abilities will be assessed using the Oxford Cognitive Screen (OCS). The OCS assesses the major cognitive domains of memory, language, number, praxis, executive functions and attention. It has been designed as a screening tool which provides a rapid assessment (approximately 15 minutes) of a patient's cognitive function. The OCS is inclusive for patients with aphasia and neglect.
Ecological Momentary Assessment App | 7 days
  This study will use a smart ecological momentary assessment delivered via a smart - phone app (smart EMA). The smart EMA samples in -the- moment data of fatigue and activity. Participants record fatigue levels (on a VAS) and contextual factors alongside every day and meaningful occupational participation from pre-defined lists. The app was developed using an iterative, user centred design and is grounded in the fatigue experiences of people with acquired brain injury, including stroke. It has been tested on participants with brain injury in the community and received good response and completion rates, with high levels of satisfaction. The participant will be prompted five times a day to record their activity and fatigue levels over a seven day period.

OTHER OUTCOMES:
Accelerometer | 7 days
  Accelerometers are portable, non - invasive wrist worn devices used to quantify physical activity with patients with a neurological condition, including stroke. Here, data can be collected in the precise moment the activity is occurring, alleviating bias. Axivity AX3 accelerometer will be worn on wrist of dominant hand over a seven day period.

CONTACTS AND LOCATIONS:
Overall Officials: Avril Dillon, BSc, Principal Investigator — Oxford Brookes University
Locations (1):
- Health and Life Sciences, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hubacher M, Calabrese P, Bassetti C, Carota A, Stocklin M, Penner IK. Assessment of post-stroke fatigue: the fatigue scale for motor and cognitive functions. Eur Neurol. 2012;67(6):377-84. doi: 10.1159/000336736. Epub 2012 May 17. PMID 22614741
- [Background] Penner IK, Raselli C, Stocklin M, Opwis K, Kappos L, Calabrese P. The Fatigue Scale for Motor and Cognitive Functions (FSMC): validation of a new instrument to assess multiple sclerosis-related fatigue. Mult Scler. 2009 Dec;15(12):1509-17. doi: 10.1177/1352458509348519. Epub 2009 Dec 7. PMID 19995840